CLINICAL TRIAL: NCT04311801
Title: Optical Coherence Tomography in Elderly Patients After Elective Orthopaedic Surgery
Brief Title: Optical Coherence Tomography (OCT) in Elderly Patients After Elective Orthopaedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk Hospital Usti nad Labem (Other)
Responsible Party: Principal Investigator, Tomas Parizek, Principal Investigator, Masaryk Hospital Usti nad Labem
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OCT
Record Dates: First submitted 2020-02-18; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Change; Retina
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OCT Arm (Experimental): Each patient underwent OCT examinations.
  Interventions: Diagnostic Test: Optical Coherence Tomography

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography — Every patient underwent OCT examination before and after surgery.

SUMMARY:
After obtaining informed consent each patient underwent OCT examination, usually one day before elective orthopaedic surgery (knee replacement). The OCT examination was repeated after the surgery. Both eyes were examined separately. After obtaining data the investigators compared the difference.

DETAILED DESCRIPTION:
Inclusion and exclusion criteria evaluated during the pre-anesthesia visit. After obtaining informed consent, patients were referred to OCT examination in the Ophthalmology clinic. The examination was performed in the 48 hours before the surgery. Between the fourth and the seventh postoperative day, the patients underwent control OCT examination. The results of OCT examinations, baseline clinical data and the data on the course of surgery and postoperative care were recorded for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Signed informed consent
* Elective operation

Exclusion Criteria:

* Age under 18
* Refusal to sign informed consent
* Non-elective operation
* Hospitalization on ICU more than 48 hours after surgery Inability to undergo OCT examination Protocol violation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Retinal changes | 4.-7. day post surgery
  Patients undergo OCT (Optical Coherence Tomography) examination of both eyes before and after the surgery.

REFERENCES:
- [Background] Roth S. Perioperative visual loss: what do we know, what can we do? Br J Anaesth. 2009 Dec;103 Suppl 1(Suppl 1):i31-40. doi: 10.1093/bja/aep295. PMID 20007988
- [Background] Gupta D, Asrani S. Macular thickness analysis for glaucoma diagnosis and management. Taiwan J Ophthalmol. 2016 Jan-Mar;6(1):3-7. doi: 10.1016/j.tjo.2016.01.003. Epub 2016 Feb 28. PMID 29018702
- [Derived] Parizek T, Skulec R, Liehneova I, Prasek P, Cerny V. No significant retinal damage induced by major orthopedic surgery - a pilot study. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2022 May;166(2):217-221. doi: 10.5507/bp.2021.022. Epub 2021 Apr 19. PMID 33885047
- See also: American Society of Anesthesiologists (ASA) classification — https://www.asahq.org/standards-and-guidelines/asa-physical-status-classification-system
- See also: OCT in clinical practice — http://eyewiki.org/Optical_Coherence_Tomography_in_Neuro-ophthalmology